CLINICAL TRIAL: NCT00883493
Title: A Randomised, Multi-Centre Study to Compare the Efficacy and Safety of Extended Release Quetiapine Fumarate (Seroquel XR TM) Tablets as Mono-Therapy or in Combination With Lithium in the Treatment of Patients With Acute Bipolar Depression
Brief Title: Efficacy and Safety of Quetiapine Versus Quetiapine Plus Lithium in Bipolar Depression
Acronym: QUALITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00055
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Acute Bipolar Depression
Keywords: Acute bipolar depression; Lithium carbonate; quetiapine fumarate; MADRS
MeSH Terms: interventions — Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapin fumarate XR (Experimental): Quetiapine XR (extended release) will be administered once daily at bedtime in oral tablet form, Day 1: 50 mg, Day 2: 100 mg, Day 3: 200 mg, Day 4 onwards: 300 mg.
  Interventions: Drug: Quetiapine fumarate XR
- Quetiapin fumarate XR+Lithium carbonate (Experimental): Quetiapine XR will be administered like monotherapy arm. Lithium will be administered twice daily from Day 1 to Day 56.
  Interventions: Drug: Quetiapine fumarate XR; Drug: Lithium carbonate

INTERVENTIONS:
Drug: Quetiapine fumarate XR — Quetiapine XR (extended release) will be administered once daily at bedtime in oral tablet form, Day 1: 50 mg, Day 2: 100 mg, Day 3: 200 mg, Day 4 onwards: 300 mg.
  Other Names: SEROQUEL XR
Drug: Lithium carbonate — Twice daily from Day 1 to Day 56. From Day 1 to Day 7, the total daily dose of lithium could be increased gradually within the dose range 300 mg/day to 1800 mg/day. From Day 8 to Day 56, the total daily dose could be adjusted from 600 to 1800 mg/day
  Other Names: LITHURIL Tb in TURKEY; LITOCARB in PERU
  Arms: Quetiapin fumarate XR+Lithium carbonate

SUMMARY:
The purpose of this study is to compare the efficacy of quetiapine fumarate monotherapy with quetiapine fumarate in combination with lithium in the treatment of a major depressive episode in patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients that meet the diagnostic criteria for bipolar disorder I and bipolar disorder II with the most recent episode depressed
* The total score of the scale that's used for the evaluation of depression (HAM-D) should be ≥20
* The total score of the scale that' used for the evaluation of mania (YMRS) should be ≤12

Exclusion Criteria:

* Patients with a current DSM-IV-TR Axis I disorder other than bipolar disorder within 6 months of enrollment. Patients who pose a current serious suicidal or homicidal risk
* Use of drugs that induce or inhibit the hepatic metabolizing enzymes within 14 days before randomisation
* Patients who are unable to discontinue all psychoactive medications, including antidepressants, antipsychotics, and mood stabilizers at least 7 days prior to randomisation and consistent with the pharmacokinetics of the drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simavi Vahip, Prof. Dr., Principal Investigator — Ege University Faculty of Medicine Psychiatry Department İzmir
Locations (24):
- Argentina (4):
  - Research Site, La Plata, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Caba
- Brazil (3):
  - Research Site, Aparecida de Goiânia, Goiás
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, São Paulo, São Paulo
- Research Site, Santiago, Chile, Chile
- Colombia (2):
  - Research Site, Medellín, Antioquia
  - Research Site, Bogota D.c, Cundinamarca
- Research Site, Guatemala City, Ciudad de Guatemala, Guatemala
- Mexico (4):
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Durango
  - Research Site, Monterrey
- Research Site, Lima, Lima Province, Peru
- Turkey (Türkiye) (7):
  - Research Site, Ankara, Turkey
  - Research Site, Elâzığ, Turkey
  - Research Site, Istanbul, Turkey
  - Research Site, Izmir, Turkey
  - Research Site, Kocaeli, Turkey
  - Research Site, Malatya, Turkey
  - Research Site, Manisa, Turkey
- Research Site, Caracas, Venezuela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject in (FSI): 22 Apr 2009, Last Subject Last Visit (LSLV): 01 Mar 2011, in 9 countries, 29 Psychiatry centres, 421 randomised participants
Pre-assignment Details: An enrollment period of up to 7 days and if applicable a wash-out period for 7-28 days depending on the medication being used, ie. antidepressants, antipsychotics and/or mood stabilizers.
Groups:
- Quetiapine XR: Quetiapine XR administered once daily in oral tablet form, Day 1: 50 mg, Day 2: 100 mg, Day 3: 200 mg, Day 4 onwards: 300 mg.
- Quatiapine XR + Lithium: Quetiapine XR administered once daily in oral tablet form, Day 1: 50 mg, Day 2: 100 mg, Day 3: 200 mg, Day 4 onwards: 300 mg. Lithium carbonate administered twice daily from Day 1 to Day 56. From Day 1 to Day 7, the total daily dose within the dose range 300 mg/day to 1800 mg/day. From Day 8 to Day 56, the total daily dose adjusted from 600 to 1800 mg/day.
Period: Overall Study
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Started | 212 | 209
Intention To Treat Analysis Population | 204 | 195
Per Protocol Analysis Population | 162 | 155
Completed | 166 | 159
Not Completed | 46 | 50
Not completed — Adverse Event | 11 | 12
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 11 | 20
Not completed — Eligibility Criteria not fullfilled | 6 | 6
Not completed — Study specific disc. criteria | 2 | 0
Not completed — Other | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium | Total
Number analyzed (Participants) | 204 | 195 | 399
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (10.8) | 39.9 (12.1) | 40.3 (11.4)
Age, Customized [Median (Full Range); unit: years] | 40 [19 to 64] | 40 [18 to 65] | 40 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 138 | 285
  Male | 57 | 57 | 114
Body weight [Mean (Standard Deviation); unit: Kilograms] — The overall number of subject the measures are reported is 398- the weight of one patient from Quatiapine XR + Lithium Arm has not been recorded at baseline.
  Kilograms | 72.8 (16.3) | 72.3 (15.4) | 72.5 (15.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score.
Description: The change of MADRS Total Score from baseline to the end of treatment was calculated by subtracting the MADRS Total Score assessed at week 8 from the baseline one (Baseline - 8 weeks).
  The MADRS is a 10-item scale that evaluates the core symptoms and cognitive features of clinical depression. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Baseline, 8 weeks
Population: The analysis population was "Per Protocol" (PP).This population included all randomized patients, classified according to medication actually received, who took study medication with not less than 75% compliance and who had a randomisation MADRS assessment and all post-randomisation MADRS assessments within pre-defined time windows at each visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
scores on a scale | 23.7 (8.4) | 24.3 (7.9)

2. Secondary Outcome: Response Rate for MADRS.
Description: Response rate defined as the percentage of patients with a ≥50% reduction from baseline in the MADRS total score to the final assessment at week 8.
  The MADRS is a 10-item scale that evaluates the core symptoms and cognitive features of clinical depression. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
percentage of participants | 93.2 (5,0) [5.0 to 6.9] | 92.9 (4,3) [4.3 to 6.2]

3. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D) Total Score.
Description: The mean change of HAM-D Total Score from baseline to the end of treatment was calculated by subtracting the HAM-D Total Score assessed at week 8 from the baseline one (Baseline - week 8).
  HAM-D is a multiple choice questionnaire used to rate the severity of a patient's major depression. It consists of 17 different items with possible scores from 0 to 4 or 0 to 2 or 0 to 6 depending on the items. Sum the total of all seventeen items gives the HAM-D Total Score, which may range from 0 (min) to 53 (max). The higher the score, the more severe the depression.
Time Frame: Baseline, 8 Weeks
Population: The analysis population was "Per Protocol" (PP).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
scores on a scale | 20.5 (7.0) | 21.0 (6.1)

4. Secondary Outcome: Change in Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The mean change in HAM-A total score from baseline to final assessment was calculated by subtracting the HAM-A Total score assessed at week 8 from the total score assessed at the baseline (baseline - week 8).
  The HAM-A is a 14-item scale that assesses anxiety symptoms of anxiety such as "anxious mood", "tension" or "fears". Each item is scored on a 5-point scale, ranging from 0=not present to 4=severe. Sum the scores from all 14 parameters gives the HAM-A Total Score which may range from 0 (min) to 56 (max).
Time Frame: baseline, 8 weeks
Population: The analysis population was "Per Protocol" (PP).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
scores on a scale | 17.5 (8.2) | 17.7 (8.2)

5. Secondary Outcome: Change in the Clinical Global Impression Severity (CGI-S) Score.
Description: The reported mean change in the CGI-S score was calculated as baseline - week 8.
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. A patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: baseline, 8 weeks
Population: The analysis population was "Per Protocol" (PP).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
scores on a scale | 3.1 (1.4) | 3.3 (1.2)

6. Secondary Outcome: Change in Young Mania Rating Scale (YMRS) Total Score.
Description: The YMRS is a rating scale to assess manic symptoms. The scale has 11 items and is based upon patient's subjective report of his or hers clinical condition over the previous 48 hours.
  The mean change in YMRS Total score reported was calculated as baseline - week 8.
  The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Time Frame: baseline, 8 weeks
Population: The analysis population was "Per Protocol" (PP).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 162 | 155
scores on a scale | 2.3 (1.8) | 2.2 (1.7)

7. Secondary Outcome: Change in the Pittsburgh Sleep Quality Index (PSQI)Total Score.
Description: The mean change in PSQI score from baseline to final assessment at week 8 was calculated as baseline - week 8.
  PSQI evaluates 7 areas of quality and pattern of sleep: sleep quality, duration getting to sleep, sleep duration, sleep adequacy, sleep disturbance, use of sleeping pill, and somnolence). Each area is rated on a scale from 0 (better) to 3 (worse) with a total score ranging from 0 to 21. Reduction in total scores are associated with better sleep quality.
Time Frame: Baseline, 8 weeks
Population: The analysis has been performed in modified Per Protocol (PP) population as this Outcome Measure was included after protocol amendment at the stage the recruitment period was already on-going.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 75 | 67
Scores on a scale | 3.7 (-20) [-20 to 21] | 5.0 (-16) [-16 to 19]

8. Secondary Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) Total Score.
Description: The mean change in (Q-LES-Q-Short Form) Total Score from baseline to week 8 was calculated by subtracting the 8 week value from baseline value (baseline - week 8).
  The Q-LES-Q-SF is a patient self assessment questionnaire consisting of 16 self-rated questions (1 being very poor - 5 very good); the first 14 will be incorporated into a total score. Higher scores indicate better quality of life.
Time Frame: baseline, 8 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 75 | 64
scores on a scale | -17.9 (12.0) [-38 to 27] | -18.8 (13.4) [-49 to 8]

9. Secondary Outcome: Change in the Sheehan Disability Scale (SDS) Total Score.
Description: The mean change in the SDS Total score from baseline to week 8 (baseline- week 8).
  Sheehan Disability Scale is a 5 item scale, with a visual analog scale evaluating work/school work, social life and family life ranging from 0 to a maximum score of 30. Each one of the 3 domains is rated from 0-10 (no impairment to most severe impairment) with evaluation of not at all (0), mild (1-3), moderate (4-6), marked (7-9) and extreme (10) disability. A total score will be calculated. A score of 30 indicates most severe impairment.
Time Frame: baseline, 8 weeks
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 76 | 66
scores on a scale | 14.4 (-3) [-3 to 30] | 14.3 (-16) [-16 to 30]

10. Secondary Outcome: Treatment Satisfaction Questionnaire (TSQ) Scores.
Description: The 14-item TAQ questionnaire evaluates the patient's overall level of satisfaction with the study medication, the effectiveness, side effects and convenience of the medication.
  Effectiveness, side effects, convenience and global satisfaction is rated on a scale of 0 being the worst and 100 being very effective, no side effects or very convenient or very satisfied. Overall satisfaction is rated over a score of 5 and 5 being the best overall satisfaction.
Time Frame: baseline, 8 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Number analyzed (Participants) | 69 | 42
Scores on a scale
  Effectivenes, baseline | 42.7 (20.2) [15.3 to 100] | 36.7 (23.7) [22.2 to 100]
  Effectivenes, week 8 | 68.7 (24.9) | 66.7 (21.8)
  Side effects, baseline | 41.7 (25.9) | 44.4 (24.9)
  Side effects, week 8 | 58.2 (26.7) | 50.4 (17.0)
  Convenience, baseline | 53.8 (21.5) | 52.8 (21.8)
  Convenience, week 8 | 73.6 (17.1) | 72.9 (17.2)
  Global satisfaction, baseline | 37.4 (26.1) | 35.0 (27.7)
  Global satisfaction, week 8 | 69.4 (19.4) | 70.7 (18.9)

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Quatiapine XR + Lithium
Serious Adverse Events (participants affected / at risk) | 5/212 | 5/209
Other Adverse Events (participants affected / at risk) | 147/212 | 149/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=212) | Quatiapine XR + Lithium (N=209)
Hospitalization due to suicide risk (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0
Appendicitis (Gastrointestinal disorders) | 1 | 0
Somnolance (Nervous system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Confusion (Nervous system disorders) | 0 | 1
Exacerbation of symptoms (Nervous system disorders) | 1 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=212) | Quatiapine XR + Lithium (N=209)
Dry mouth (Nervous system disorders) | 50 | 47
Somnolance (Nervous system disorders) | 46 | 49
Headache (Nervous system disorders) | 28 | 25
Anxiety (Nervous system disorders) | 21 | 14
Constipation (Gastrointestinal disorders) | 20 | 17
Dizziness (Nervous system disorders) | 16 | 32
Diarrhea (Gastrointestinal disorders) | 14 | 13
Nausea (Gastrointestinal disorders) | 14 | 29
Increased appetite (Nervous system disorders) | 13 | 5
Tremor (Nervous system disorders) | 11 | 28
Sedation (Nervous system disorders) | 9 | 11
Weight gain (General disorders) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other